# **Informed Consent Form (ICF)**

The Effects of Weight Science and Nutrition Education on Weight Control Beliefs, Body Image, Self-Esteem and Eating Patterns in Undergraduate Dieters

Unique Protocol ID #19334

November 4<sup>th</sup>, 2025





## Consent Form

Title of Study: The Effects of Weight Science and Nutrition Education on Weight Control Beliefs, Body Image, Self-Esteem and Eating Patterns in Undergraduate Dieters

Locally Responsible Investigator and Principal Investigator, Department/Hospital/Institution: Dr. Keisha Gobin, Eating Disorders Clinic, St. Joseph's Healthcare Hamilton

Student Investigators, Department/Hospital/Institution: Mindy Tat, McMaster University; Sarah Potter, McMaster University

You are being invited to participate in a research study conducted by Mindy Tat as an undergraduate student at McMaster University under the supervision of Dr. Keisha Gobin.

In order to decide whether or not you want to be a part of this research study, you should understand what is involved and the potential risks and benefits. This form gives detailed information about the research study. If you have any questions about the study, please contact Dr. Keisha Gobin at <a href="kgobin@stjosham.on.ca">kgobin@stjosham.on.ca</a>. Once you understand the study, you will be asked to sign this form if you wish to participate. Please take your time to make your decision.

Neither Dr. Gobin nor her fellow researchers have any conflict of interest to declare in conducting this study.

#### WHAT IS THE PURPOSE OF THIS STUDY?

I, Mindy Tat, am carrying out this study as part of the requirements for my Honours Bachelor of Science Degree. The purpose of this study is to evaluate the effects of different types of education on your beliefs and attitudes about weight and healthy living, and how these in turn affect things like your body satisfaction and self-esteem.

#### WHAT WILL MY RESPONSIBILITIES BE IF I TAKE PART IN THE STUDY?

If you agree to participate in the study, you will be asked to do the following things:

You will be asked to watch 2 videos and answer a series of online questionnaires. The first set of questionnaires will ask you information about your gender, ethnicity, physical activity levels, eating patterns, body image, the intent to diet, beliefs about weight, self-esteem, and behaviours related to body image. After these questionnaires you will watch two educational videos related to living a healthy lifestyle. Finally, you will complete a second set of questionnaires about eating patterns, body image, the intent to diet, beliefs about weight, self-esteem, and behaviours related to body image. When you have completed the questions, you will press 'Submit' at the bottom of the page to complete your participation in the study. At that time, a list of resources available through McMaster University will be available to you, for your reference and/or use. This entire process should take no more than 2 hours.

Please note that by participating in this study, you do not give up any rights to which you may be entitled under the law.

### WHAT ARE THE POSSIBLE RISKS AND DISCOMFORTS?

The risks involved in this study are minimal; however, it is possible that you may feel uncomfortable or anxious when filling out some of the items in the questionnaires. We encourage you to fill out the questionnaires as completely and honestly as possible. However, you do not need to answer any question you do not wish to answer. You may leave those questions blank. You may withdraw from the study at any time by simply closing the questionnaire window and leaving the room. You will not be penalized for leaving questions blank or withdrawing from the study. If after completing the questionnaire you feel that you would like to speak to someone about any concerns you might have about your eating, activity, or thoughts about yourself, we have provided you with counselling resources that you may wish to contact. Your answers on the questionnaires will be deleted after study completion, de-identified, and exported for long-term storage in a secure server at St. Joseph's Healthcare Hamilton, which will ensure that your responses will be kept entirely private.

Because this study involves completing questionnaires online, there is a small risk of a privacy breach. Although all reasonable safeguards are in place to protect your information, absolute security cannot be guaranteed. By choosing to participate, you acknowledge and consent to this potential risk. If a privacy breach involving your identifiable information were to occur, the research team will notify you as soon as possible, provide information about the nature of the breach, and explain any steps being taken to address it.

#### HOW MANY PEOPLE WILL BE IN THIS STUDY?

We plan to collect data between January 2026 and August 2026, and we expect that the total number of people who participate in the study will be at least or approximately 150.

#### WHAT ARE THE POSSIBLE BENEFITS FOR ME AND/OR FOR SOCIETY?

We cannot promise any personal benefits to you from your participation in this study. However, you may benefit from the knowledge you retain from the educational videos as they pertain to weight science, healthy eating, and sleep. Your participation in this study will contribute to general scientific knowledge related to the impact of education on weight control beliefs and eating pathology. There are no medical benefits to you from your taking part in this study.

#### WHAT INFORMATION WILL BE KEPT PRIVATE?

All identifiable, coded, and de-identified study data will be collected and temporarily held through McMaster's secure REDCap system, which is password-protected and accessible only to authorized McMaster and study personnel. After data collection is complete, your responses will be exported and permanently deleted from McMaster's REDCap and moved to a secure, password-protected electronic system in the research laboratory at St. Joseph's Healthcare Hamilton (SJHH).

Your data will not be shared with anyone except with your consent or as required by law. All personal information such as your name, email address, and gender will be removed from the data and will be replaced with a number. A list linking the number with your name will be kept in a secure place, separate from your data. The data, with identifying information removed will be securely stored in a password-protected electronic system in the research laboratory. Your study responses and the list linking your study number with your name will be deleted from REDCap and the password-protected electronic system in the research laboratory in 10 years.

For the purpose of ensuring proper monitoring of the research study, it is possible that representatives of the Hamilton Integrated REB (HiREB), this institution, and affiliated sites may consult your original research data to check that the information collected for the study is correct and follows proper laws and guidelines. By participating in this study, you authorize such access.

If the results of the study are published, your name will not be used and no information that discloses your identity will be released or published without your specific consent to the disclosure.

#### CAN PARTICIPATION IN THE STUDY END EARLY?

If you volunteer to be in this study, you may withdraw at any time and for any reason. If you decide to withdraw from the study, there will be no consequences to you. If you decide to withdraw from the study, you will still be compensated with partial course credit. In cases of withdrawal, all data will be destroyed unless you indicate otherwise. You are able to withdraw your data up until September 15th, 2026, when we expect to submit a manuscript that details the findings of the study. You may also refuse to answer any questions you do not what to answer and still remain in the study.

To withdraw from the study, exit the questionnaire and contact the Student Investigator, Mindy Tat via email at tatm@mcmaster.ca, or in person during the allotted study time. She will ensure that any data you have provided is destroyed.

#### WILL I BE PAID TO PARTICIPATE IN THIS STUDY?

projectredcap.org

There is no monetary payment available for participating in this study. You will be compensated with partial course credit for your participation.

## IF I HAVE ANY QUESTIONS OR PROBLEMS, WHOM CAN I CALL?

If you have any questions about the research now or later, you can call Dr. Keisha Gobin at 905-522-1155 extension 34093.



2025/11/04 - V.2 projectredcap.org

| | CONSENT STATEMENT | | |
|---|---|---|---|
| 1) | 1) Participant: I have read the preceding information thoroughly. I have had an opportunity to ask questions and of my questions have been answered to my satisfaction. I agree to participate in this study. I understand that I v receive a signed copy of this form. | | |
| | ○Yes | | |
| | If you would like to discuss the study in more detail before signing, please 34093 or email her at kgobin@stjoes.ca. | contact Dr. Keisha Gobin at 905-5 | 22-1155 extension |
| 2) | 2) First Name: | | |
| 3) | 3) Last Name: | | |
| 4) | 4) Signature: | | |
| | | | <u></u> |
| 5) | 5) Date: | | - |
| | Consent form reviewed by: | | |
| | (researcher's signature) | | |
| 6) | 1) First Name: | | |
| 7) | 2) Last Name: | | |
| 8) | 3) Signature: | | |

This study has been reviewed by the Hamilton Integrated Research Ethics Board (HIREB). The HIREB is responsible for ensuring that participants are informed of the risks associated with the research, and that participants are free to decide if participation is right for them. If you have any questions about your rights as a research participant, please call the Office of the Chair, Hamilton Integrated Research Ethics Board at  $905.521.2100 \times 42013$ .

Consent Form Version Number and Date: Version 2 -

November 4, 2025

4) Date:

Protocol Number and Version: #19334, 2.0

**₹EDCap**®